CLINICAL TRIAL: NCT04066946
Title: Study for the Effects of Microcurrent Therapy on the Prevention and Healing of Brachioplasty Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organisation for Burns, Scar Aftercare and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP0020-201901-MCU
Record Dates: First submitted 2019-08-16; First posted 2019-08-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-11

CONDITIONS: Cicatrix
Keywords: scar; arm; brachioplasty; microcurrent; interventional study
MeSH Terms: conditions — Cicatrix | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single centre, two-arm, single blinded randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 = Intervention group (Experimental): Standard of care (hydration + silicone gel sheet) + Microcurrent
  Interventions: Device: Microcurrent therapy; Other: Standard of care
- Group 2 = Control Group (Active Comparator): Standard of care (hydration + silicone gel sheet)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Microcurrent therapy — Micro current therapy is a therapy to treat humans / animals using electric current with amperages flowing in the μA range. The device offers 2 treatment methods: manual treatment, which requires manual input corresponding to the mentioned parameters, and automatic treatment which, depending on the clinical picture and the currently measured resistance between the electrodes, allows the device to automatically change the mentioned parameters. For this study the investigators use an automatic treatment with predefined settings. This automatic programme consists of a variation of 20 different frequency settings during 17 minutes. This programme is repeated one time which leads to a total treatment time of 34 minutes. The intensity setting for the treatment is between 200 and 350 µA. The treatment is applied 5x per week in the first 6 weeks. The treatment is stopped after six weeks.
  Arms: Group 1 = Intervention group
Other: Standard of care — Standard of Care consists of:
  During the first two weeks:
  * Histoacryl glue to close the surgical incisions.
  * Suture strips to keep the wound closed.
  * Isobetadine Dermicum as anti-septic treatment
  * Dry wound dressings during the first 2 weeks.
  * Tubigrip
  From two weeks until three months:
  • Hydration with hydrating crème 2x per day (not within 4 hours before microcurrent treatment.
  From three months onwards:
  • Silicone gel sheet.

SUMMARY:
Prospective, single-centre two-arm randomized controlled trial. Both groups receive standard wound care + hydration. The intervention group also receives microcurrent therapy. Patients with surgical incisions from bilateral Brachioplasty procedures will be included in this study. One arm will be randomized in the intervention group and one arm in the control group. Objective and subjective outcomes are registered. The aim of this study is to investigate whether the outcomes of the patients of the intervention group differ significantly from the patients in the control group.

DETAILED DESCRIPTION:
Study procedures:

Description of the clinical-investigation-related procedures in order of occurrence.

Measurements will be carried out at the following time-points:

* 15 days after surgery
* 90 days after surgery
* 180 days after surgery

Measurement procedures:

All patients will respect a 30 minute acclimatisation period in the measurement room with standardised room temperature (20-22°C) and relative humidity (40-50%). Patients will be asked to remove their silicones and pressure garments the evening before the actual measurement. The scar site used for testing is marked with a circular adhesive marking with a diameter of 30 mm. A picture is taken to establish the location. The following optimal patient position is recommended. For measurements on forearms and upper arms a seated position with the arm on a (massage) table.

Order of occurrence:

1. Intake questionnaire
2. Digital photographs
3. Patient and Observer Scar Assessment
4. Colour measurement
5. Hydration measurement
6. Elasticity measurement
7. Quality of Life questionnaires

Intake questionnaire Patient will be asked to fill out an intake form with all relevant information for the study. This will include age, body weight, gender, ethnicity, date of surgery, smoking, scar revision or initial treatment,

Digital Photographs A digital photograph will be taken from the patient's face and/or neck. This photograph will be taken from a standardised distance.

Patient and Observer reported Scar Assessment Scale (PSAS-OSAS) The POSAS aims to measure scar quality. Current developments in scar treatment necessitate reliable and valid scar assessment tools. The POSAS is a comprehensive scale that is designed for the evaluation of all types of scars by professionals and patients. The Patient Scale gives the POSAS an important extra dimension because the patient's opinion is mandatory for a complete scar evaluation. When patients indicated may update their opinion without having to visit the hospital. This can be achieved at their convenience by internet or e-mail.

Clinimetric studies support the use of the POSAS for subjective scar evaluation. The first publication on the POSAS (Version 1.0) was in 2004. With one extra item for the Observer Scale and minor textual modifications POSASv2.0 was tested on linear scars and published in 2005.

The POSASv2.0 consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores' of the Patient and Observer Scale. Furthermore category boxes are available to score nominal parameters (e.g. type of colour). Moreover, the patient and observer also score their 'Overall Opinion'.

Colour measurement with Mexameter® Light is generated by a source lamp and is dispersed into its constituent wavelengths in a monochromator which results in a narrow band of the dispersed spectrum passing from the exit slit of the device. Suitable optics is used to lead this light, of a narrow wavelength band, to the sample being measured. A sample with an UV/Visible chromophore sample absorbs a certain amount of light and a suitable detector in the spectrophotometer detects the remaining light. The Beer-Lambert law is then applied to determine the concentration of the remaining light in the sample at a specific wavelength. The most commonly used wavelengths are 568 nm (green), 660 nm (red) and 880 nm (infrared). A melanin index can be computed from the results of red and infrared wavelengths and an erythema index is calculated from the results of green and red wavelength. Draaijers et al. stated that it is easier to understand the meaning of the erythema and the melanin index than the L*a*b* values.

Hydration measurements with Corneometer CM825 The measuring principle is based on the capacitance method. Technical description of this type of instrument and its use has been published by many authors. Both probes (analog and digital) contain an inter-digital grid of gold electrodes, covered by a low dielectric vitrified material. A resonating system in the instrument detects the frequency shift of the oscillating system related to the capacitance (and hence hydration) of the biomaterial in contact with the probe. Unlike other instruments, there is no direct galvanic contact between the electrodes of the Corneometer and the skin surface. To enable a constant pressure of the probe on the skin surface a spring system is incorporated. According to the manufacturer the pressure of the old analog probe is in the range of 1.1-1.8 N, the new digital probe operates at a lower pressure (about 1 N or less). The Corneometer is factory-calibrated using an in vitro method. The principle of this in vitro calibration system developed by Courage-Khazaka for the Corneometer is based on the use of a C-K reference filter pad soaked with a calibration solution (saturated NaCl solution in water). With this impregnated filter pad a maximal hydration value of 120 ± 5 AU can be attained. When covering the surface of the impregnated pad with one layer of a very thin polyurethane foil, a hydration value of about 20 ± 5 AU should be obtained.

Elasticity measurements with Cutometer® MPA580 The Cutometer® is designed to measure elasticity of the upper skin layer using negative pressure which mechanically deforms the skin. The measuring principle is based on the suction method. Negative pressure is created in the device and the skin is drawn into the aperture of the probe and released again after a defined time. Inside the probe the penetration depth is determined by a non-contact optical measuring system. This optical measuring system consists of a light source and a light receptor and two prisms facing each other that project the light from transmitter to receptor. The light intensity varies due to the penetration depth of the skin. The resistance of the skin to the negative pressure (firmness) and its ability to return to its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time during the measurement. This measurement principle allows data collection on the elastic and mechanical properties of skin surface and enables objective quantification of skin aging. The Cutometer® measures the vertical deformation of the skin in millimetres when the skin is pulled by means of a controlled vacuum into the circular aperture of the probe.

Quality of Life Questionnaires

EQ5D:

The EQ-5D was developed by the EuroQol Group, an international, cross-disciplinary group that was set up in 1987 to investigate issues related to the evaluation of health. It has been translated to more than 60 languages, is used worldwide and has previously been used in Swedish population. The reliability and validity of EQ-5D have been documented, both in general and in burns-specific population.

The EQ-5D descriptive system encompasses five questions covering five dimensions: mobility, self-care, usual activities, pain and anxiety/depression. For each dimension, respondents value their health by reporting whether they are experiencing 1 = ''none'', 2 = ''moderate'' or 3 = ''extreme problems''. A unique EQ-5D health state is defined by combining the responses (1, 2 or 3) on each of the five dimensions. The EQ VAS is a vertical 20-cm line graded from 0 = ''worst possible health state'' to 100 = ''best possible health state'', on which the respondent is asked to mark his or her own current state of health. The EQ-5D health state can also be converted into a weighted index. The conversion into the index is based on norm values obtained in population-based enquiries. The EQ-5D index ranges from 0.594 = ''death or worse than death'' to 1 = ''full health''.

Dermatology Life Quality Index:

The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above.

There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life)

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be between 18 and 75 years old.
* Having received surgical treatment, more specific bilateral brachioplasty.

Exclusion Criteria:

* Subjects who have an implanted or other electrical stimulatory device such as pacemakers, or any other implanted electronic nerve, muscle or tissue stimulation.
* Subjects with implanted hearing aids.
* Subjects with a history of seizures, epilepsy.
* Women who are pregnant at the time of enrolment
* Central neurological conditions
* Peripheral paralysis
* Patients with diabetes mellitus
* Subjects unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Assessing the change of POSAS Patient Scale Total Sum of Scores | At baseline (15 days after surgery) - 180 days after surgery.
  The POSAS Patient Scale contains six items (pain, itch, colour, thickness, pliability, texture) that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores'.

SECONDARY OUTCOMES:
POSAS Observer Scale Total Sum of Scores | At visit 1 (15 days after surgery) - at visit 2 (90 days after surgery) - at visit 3 (180 days after surgery)
  The POSAS Observer Scale contains six items (vascularity, pigmentation, colour, thickness, pliability, surface) that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores'.
Colour measurement with MexaMeter | At visit 1 (15 days after surgery) - at visit 2 (90 days after surgery) - at visit 3 (180 days after surgery)
  Light is generated by a source lamp and is dispersed into its constituent wavelengths in a monochromator which results in a narrow band of the dispersed spectrum passing from the exit slit of the device. Suitable optics is used to lead this light, of a narrow wavelength band, to the sample being measured. A sample with an UV/Visible chromophore sample absorbs a certain amount of light and a suitable detector in the spectrophotometer detects the remaining light. The Beer-Lambert law is then applied to determine the concentration of the remaining light in the sample at a specific wavelength. The most commonly used wavelengths are 568 nm (green), 660 nm (red) and 880 nm (infrared). A melanin index can be computed from the results of red and infrared wavelengths and an erythema index is calculated from the results of green and red wavelength. Draaijers et al. stated that it is easier to understand the meaning of the erythema and the melanin index than the L*a*b* values.
Elasticity measurement with Cutometer | At visit 1 (15 days after surgery) - at visit 2 (90 days after surgery) - at visit 3 (180 days after surgery)
  The Cutometer® is designed to measure elasticity of the upper skin layer using negative pressure which mechanically deforms the skin. The measuring principle is based on the suction method. Negative pressure is created in the device and the skin is drawn into the aperture of the probe and released again after a defined time. Inside the probe the penetration depth is determined by a non-contact optical measuring system. This measurement principle allows data collection on the elastic and mechanical properties of skin surface and enables objective quantification of skin aging. The Cutometer® measures the vertical deformation of the skin in millimetres when the skin is pulled by means of a controlled vacuum into the circular aperture of the probe.
Generic assessment of Quality of Life with EQ5D | At visit 1 (15 days after surgery) - at visit 2 (90 days after surgery) - at visit 3 (180 days after surgery)
  The EQ-5D descriptive system encompasses five questions covering five dimensions: mobility, self-care, usual activities, pain and anxiety/depression. For each dimension, respondents value their health by reporting whether they are experiencing 1 = ''none'', 2 = ''moderate'' or 3 = ''extreme problems''. A unique EQ-5D health state is defined by combining the responses (1, 2 or 3) on each of the five dimensions. The EQ VAS is a vertical 20-cm line graded from 0 = ''worst possible health state'' to 100 = ''best possible health state'', on which the respondent is asked to mark his or her own current state of health. The EQ-5D health state can also be converted into a weighted index. The conversion into the index is based on norm values obtained in population-based enquiries. The EQ-5D index ranges from 0.594 = ''death or worse than death'' to 1 = ''full health''.
Disease specific assessment of Quality of Life with DLQI | At visit 1 (15 days after surgery) - at visit 2 (90 days after surgery) - at visit 3 (180 days after surgery)
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above.
  There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Moortgat, Study Director — OSCARE npo
Locations (1):
- Organisation for burns, scar after-care and research, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No